CLINICAL TRIAL: NCT03415750
Title: A Single-center,Randomized,Open-label,12 Months Study,2 Parallel Group to Compare the Efficacy of Everolimus Combination + Tacrolimus in Regression of Left Ventricular Hypertrophy vs Tacrolimus + MMF in Renal Transplant Patients
Brief Title: Everolimus and Tacrolimus Combination for Regression of Left Ventricular Hypertrophy in Renal Transplants
Acronym: ENHVIE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edoardo Melilli (Other)
Responsible Party: Sponsor-Investigator, Edoardo Melilli, Principal Investigator MD, Hospital Universitari de Bellvitge
Organization: Hospital Universitari de Bellvitge (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ENHVIE
Record Dates: First submitted 2016-11-17; First posted 2018-01-30 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2021-01

CONDITIONS: Hypertrophy, Left Ventricular
Keywords: Renal transplant
MeSH Terms: conditions — Hypertrophy, Left Ventricular | interventions — Everolimus; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Everolimus arm (Experimental): Patients will be converted from Tacrolimus + Mycophenolate mofetil to Everolimus + Tacrolimus 'Conversion from Mycophenolate mofetil to Everolimus'
  Interventions: Drug: Everolimus; Drug: Tacrolimus
- Mycophenolate arm (Active Comparator): Patients will remain in Tacrolimus + Mycophenolate mofetil combination
  Interventions: Drug: Mycophenolate mofetil; Drug: Tacrolimus

INTERVENTIONS:
Drug: Everolimus — Conversion from Mycophenolate mofetil to Everolimus
  Other Names: Certican
  Arms: Everolimus arm
Drug: Mycophenolate mofetil — Patients will remain in Tacrolimus + Mycophenolate mofetil
  Other Names: Cellcept
  Arms: Mycophenolate arm
Drug: Tacrolimus
  Other Names: Prograf

SUMMARY:
Clinical study with two parallel group to compare the efficacy of everolimus combination + tacrolimus in regression of left ventricular hypertrophy vs tacrolimus + mycophenolate mofetil in renal transplant patients in the maintenance phase.

DETAILED DESCRIPTION:
A single-center, randomized, open-label, 12 months study, with two parallel group to compare the efficacy of everolimus combination + tacrolimus in regression of left ventricular hypertrophy vs tacrolimus + mycophenolate mofetil in renal transplant patients in the maintenance phase.

ELIGIBILITY:
Inclusion Criteria:

* Patient's signed informed consent prior to any study-related procedure.
* Adult patients (> 18 years), renal transplant recipients of more than 1 year of evolution.
* Patients receiving maintenance immunosuppression with tacrolimus delayed release (Envarsus®) and MMF / MPA.
* Patients with Left Ventricular Hypertrophy detected by Cardio-NMR.
* Subjects with glomerular filtration rate >30 ml/min (calculated by CKD-EPI) and stable in the last two analytical determinations (variation <20%).
* No known contraindications to the use of Mtor inhibitors (previous intolerance, deep vein thrombosis , pulmonary embolism, proteinuria > 0.5 g/day)
* Patients with Hb levels ≥ 11 gr/dl.
* Patients with blood pressure <140/90 mmHg in the hospital visits or <135/85 mmHg at home.

Exclusion Criteria:

* Patient's signed informed consent prior to any study-related procedure.
* Adult patients (> 18 years), renal transplant recipients of more than 1 year of evolution.
* Patients receiving maintenance immunosuppression with tacrolimus delayed release (Envarsus®) and MMF / MPA.
* Patients with Left Ventricular Hypertrophy detected by Cardio-NMR.
* Subjects with glomerular filtration rate >30 ml/min (calculated by CKD-EPI) and stable in the last two analytical determinations (variation <20%).
* No known contraindications to the use of Mtor inhibitors (previous intolerance, deep vein thrombosis , pulmonary embolism, proteinuria > 0.5 g/day)
* Patients with Hb levels ≥ 11 gr/dl.
* Patients with blood pressure <140/90 mmHg in the hospital visits or <135/85 mmHg at home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Reduction of Left Ventricular Hypertrophy | 12 months
  Reduction of Left Ventricular Hypertrophy more or equal than 10 g/m2 in the study group compared to control group at 12 months. Regression of LVH is defined as a decrease of 10 g/m2 compared to baseline value. Cardio nuclear magnetic resonance will be performed to evaluate left ventricular hypertrophy

CONTACTS AND LOCATIONS:
Overall Officials: Edoardo Melilli, MD, Principal Investigator — Hospital Universitari de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No